CLINICAL TRIAL: NCT01086787
Title: Paracrine Mechanisms of Bone Marrow Stem Cell Signalling in Chronic Heart Failure
Acronym: BM-CHF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: R.A. de Boer, MD, PhD, University Medical Center Groningen
Other Study IDs: WTR-ECG-5
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-03

CONDITIONS: Heart Failure
Keywords: Heart failure; Bone marrow; Bone marrow mononuclear cells; Surgery; Orthopedic surgery; Cardiac surgery
MeSH Terms: conditions — Heart Failure | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, white cells, urine, bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non heart failure patients: Patients without heart failure undergoing open chest surgery
  Interventions: Other: Surgery
- Orthopedic patients: Patients without heart failure undergoing orthopedic surgery
  Interventions: Other: Surgery
- Heart failure patients: Patients with heart failure undergoing open chest surgery.
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Surgery — Patients undergoing surgery for either cardiac surgery or orthopedic surgery

SUMMARY:
The investigators hypothesize that chronic heart failure is associated with a general stem cell dysfunction, which translates into reduced paracrine function of adult stem cells from patients with chronic heart failure as compared to patients with preserved systolic function.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

1. Before any study-specific procedures, the appropriate written informed consent must be obtained.
2. Male and female older than 18 years of age.

   For the cardiac patients:
3. Being accepted for cardiothoracic surgery with the use of open chest surgery
4. A known left ventricular ejection fraction, either assessed by echocardiography, MUGA or MRI. If LVEF <40% a subject will be assigned to the chronic heart failure group, if LVEF >40% a subject will be assigned to the control group.

   For the non-cardiac patients:
5. Accepted for orthopedic surgery (e.g. total hip replacement) at the department of orthopedic surgery.

Exclusion Criteria:

1. An unstable medical condition, defined as having been hospitalized for a non-cardiac condition within 4 weeks of screening, or otherwise unstable in the judgment of the investigator (e.g. at risk of complications or adverse events unrelated to study participation).
2. Younger than 18 years of age.
3. Clinical history of chronic kidney disease (at any point prior to registration).
4. Any known hepatic disease.
5. Recent (within 3 months) history of alcohol or illicit drug abuse disorder, based on self-report.
6. Clinically significant abnormality in chemistry, hematology, or urinalysis parameters performed within the screening period.
7. Participation in any investigational device or drug trial(s) or receiving investigational agent(s) within 30 days.
8. Any condition (e.g. psychiatric illness, etc.) or situation that, in the investigator's opinion, could put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
9. Legally incompetent adults, for which reason what so ever.

   For the non-cardiac patients:
10. A known history of cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Man and woman, undergoing cardiothoracic surgery, older than 18 years of age, with and without preserved left ventricular ejection fraction (LVEF <40% and >40%). Controls are man and women, older than 18 years of age, scheduled for orthopaedic surgery without a history of cardiac disease.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Paracrine properties of bone marrow cells from patients with heart failure | 1 day
  To compare the paracrine properties of bone marrow-derived stem cells harvested from patients suffering chronic heart failure vs healthy subjects. In particular, we aim to determine if the cytoprotective, pro-angiogenic and anti-fibrotic effects mediated by bone marrow stem cells of heart failure patients are similar to those from healthy patients.

SECONDARY OUTCOMES:
To study preconditioning of different bone marrow stem cells with different cytokines | 1 day
To study in detail the temporal and spatial expression of paracrine factors in bone marrow stem cells in vitro, and to study the differences between bone marrow stem cells from patients with and without chronic heart failure | 1 day
To evaluate potential molecular mechanisms involved | 1 day
To find mechanisms to enhance expansion of different bone marrow stem cells in vitro | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: W. T. Ruifrok, MD, Principal Investigator — University Medical Center Groningen; R. A. de Boer, MD, PhD, Study Director — University Medical Center Groningen; W. H. van Gilst, PhD, Study Chair — University Medical Center Groningen; M. Gnecchi, MD, PhD, Study Director — University of Pavia; L. Kleijn, MD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Department of Heart, Blood and Lung , University of Pavia, Pavia, Italy
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands